CLINICAL TRIAL: NCT05850104
Title: Comparison of Classical Prosthesis and Silicone Prosthesis in Patients With Chopart Amputation
Brief Title: Comparison of Classical Prosthesis and Silicone Prosthesis
Status: Completed | Type: Observational
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Associate professor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: 38
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Traumatic Amputation
Keywords: amputation; chopart; satisfaction
MeSH Terms: conditions — Amputation, Traumatic; Personal Satisfaction | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- classical prosthesis group: the effects of classical Chopart prosthesis on socket comfort, satisfaction level and quality of life in patients with unilateral Chopart amputation
  Interventions: Other: the effects of classical Chopart prosthesis on socket comfort, satisfaction level and quality of life in patients with unilateral Chopart amputation.
- silicone prosthesis group: the effects of silicone prosthesis on socket comfort, satisfaction level and quality of life in patients with unilateral Chopart amputation
  Interventions: Other: the effects of silicone prosthesis on socket comfort, satisfaction level and quality of life in patients with unilateral Chopart amputation.

INTERVENTIONS:
Other: the effects of classical Chopart prosthesis on socket comfort, satisfaction level and quality of life in patients with unilateral Chopart amputation. — the effects of classical Chopart prosthesis and silicone prosthesis on socket comfort, satisfaction level and quality of life in patients with unilateral Chopart amputation.
  Groups: classical prosthesis group
Other: the effects of silicone prosthesis on socket comfort, satisfaction level and quality of life in patients with unilateral Chopart amputation. — the effects of silicone prosthesis on socket comfort, satisfaction level and quality of life in patients with unilateral Chopart amputation.
  Groups: silicone prosthesis group

SUMMARY:
The purpose of this study is to investigate the effects of classical Chopart prosthesis and silicone prosthesis on socket comfort, satisfaction level and quality of life in patients with unilateral Chopart amputation.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effects of classical Chopart prosthesis and silicone prosthesis on socket comfort, satisfaction level and quality of life in patients with unilateral Chopart amputation.

This study will be useful for prescribing the appropriate prosthesis in patients with Chopart amputation.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-65
* Having a unilateral traumatic Chopart amputation
* To have completed prosthesis training
* Using prosthesis for at least 6 hours a day
* Being at K3-K4 activity level

Exclusion Criteria:

* Bilateral lower extremity amputation
* Presence of wound on stump
* Presence of neurological, cardiovascular, and pulmonary disease that may affect walking performance

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 24 patients with unilateral Chopart amputation
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2023-05-24 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | through study completion, an average of one and a half months
  All patients will mark the severity of residual limb pain, sound limb pain and low back pain on a Visual Analogue Scale (VAS; from 0 (no pain) to 10 (worst pain)). The socket system, prosthetic foot and overall prosthesis satisfaction will be evaluated with a 10-point VAS (from 0 (absolutely dissatisfied) to 10 (absolutely satisfied)).
Short Form 36 (SF-36) | through study completion, an average of one and a half months
  The QoL of each patient will be assessed using the Short Form 36 (SF-36). The validity and reliability of the Turkish version of SF-36 has been demonstrated. SF-36 consists of 36 questions on eight different subscales that include physical functioning, role limitations due to physical health problems, bodily pain, general health perceptions, energy and fatigue, vitality, social functioning, role limitations due to emotional problems and general mental health. Each subscale of SF-36 is scored between 0 and 100, and higher scores illustrate better QoL.
Locomotor capacity index | through study completion, an average of one month
  The Locomotor Capabilities Index (LCI) is a validated measure of lower-limb amputees' ability to perform activities with prosthesis. The total LCI score is the sum of the item scores and can range from 0 (worst) to 30 (best).
Likert scale | through study completion, an average of one month
  Level of difficulty experienced during walking on straight road, walking uneven road, ascending stairs, descending stairs, ascending ramps and descending ramps will be recorded on a 5-point Likert scale ((1) very easy, (2) easy , (3) neutral, (4) difficult, (5) very difficult).

CONTACTS AND LOCATIONS:
Overall Officials: Merve Örücü Atar, MD, Principal Investigator — associate professor
Locations (1):
- Ankara Gaziler Physical Medicine and Rehabilitation Education and Research Hospital, Ankara, Turkey (Türkiye)